CLINICAL TRIAL: NCT02081950
Title: A Single-Dose Study to Examine the Within Subject Variability of Clexane® (80 mg) s.c. in Healthy Adult Subjects Under Fasting Conditions
Brief Title: A Single-Dose Trial to Examine the Within Subject Variability of Clexane® in Healthy Adults Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chemi S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ENOXA/13/1
Record Dates: First submitted 2014-03-06; First posted 2014-03-07 (Estimated); Results first posted 2020-09-29 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-10

CONDITIONS: Clexane is Administered to Healthy Volunteers
Keywords: enoxaparin sodium
MeSH Terms: interventions — enoxaparin sodium; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enoxaparin sodium (Experimental): Enoxaparin sodium (80mg) is administered subcutaneously as a single dose, in 2 periods.
  Interventions: Biological: Enoxaparin sodium

INTERVENTIONS:
Biological: Enoxaparin sodium — comparison of 2 different administration of drug
  Other Names: Clexane

SUMMARY:
Primary: To examine the within subject variability of Clexane (80 mg) in healthy male and female volunteers administered subcutaneously (s.c.) as a single dose, in two periods, under fasting conditions.

Secondary: To monitor safety during the Treatment Periods.

DETAILED DESCRIPTION:
This was a pilot, open-label study to evaluate the PK of enoxaparin following s.c. administrations of 80 mg Clexane, on 2 different occasions, in 14 healthy adult subjects.

The study comprised a Screening Visit and 2 Treatment Periods (1 and 2). Screening (Day -14 to Day -1): Screening assessments were carried out within 14 days before administration of the first dose of Clexane. Eligible subjects were asked to return for Treatment Period 1.

Treatment Periods 1 and 2 (Day 0 to Day 26): Eligible subjects received two doses of s.c. Clexane over 2 Treatment Periods (1 dose/period). Final confirmation of eligibility was made prior to dosing during Treatment Period 1. Confirmation of ongoing eligibility was made prior to dosing during Treatment Period 2.

Each Treatment Period was of 2 days duration, from the afternoon before dosing (Day 0) until 36 hours (h) post-dose (evening of Day 2). During each Treatment Period, subjects resided at the Clinical Unit. Study drug was administered on the morning of Day 1 following an overnight fast. Pharmacokinetic (PK) samples were collected pre-dose and up to 36 h post-dose (x14 samples) for the measurement of enoxaparin. Safety was also evaluated at specified times throughout the study. There were at least 7 days between each dose administration. The Post-Study Follow-Up was conducted on Day 2 of Treatment Period 2 after completion of the 36 h PK blood sampling and vital sign check.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteer between 18 and 55 years of age.
* Female subject of child bearing potential with a negative pregnancy test at the Screening Visit and willing to use 2 effective methods of contraception from Day 1 until 3 months afterwards.
* Subject with no clinically significant abnormal serum biochemistry, haematology, coagulation factors and urine examination values within 14 days of the first dose.

Exclusion Criteria:

* Female subject with weight < 45 kg or male subject with weight < 57 kg.
* Subject with clinically relevant abnormal physical findings which could interfere with the objective of the study.
* Subject with clinically relevant abnormal laboratory values indicative of physical illness; Hemoglobin <13 g/dL; Absolute platelet count below 100 x 109/L.
* Subject with hypersensitivity or idiosyncratic reaction to enoxaparin and/or low molecular weight heparins, and/or pork products.
* Subject with a relevant history or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease. In addition, history or presence of: alcoholism or drug abuse within the past year; clotting disorders; gastric or duodenal ulcers; hypertension; retinopathy; deep venous thrombosis; pulmonary embolism; GI bleeding.
* Subject with any clinically significant illness within 4 weeks prior to dosing.
* Subject with recent use of NSAID and/or aspirin (within 4 weeks of first dose) or the use of any pharmacological agents known to significantly induce or inhibit drug-metabolizing enzymes within 30 days of the first dose. No subject may take any antibiotic agent known to interfere with intestinal microflora within 30 days of the first dose. Subjects with any medical condition requiring regular treatment with prescription drugs.
* Subject with recent severe trauma, surgery (eye surgery), and/or lumbar puncture;
* Female subject who was pregnant or lactating.
* Subject who was a vegetarian.
* Subject who, through completion of the study, would have donated in excess of 500 mL of blood and/or plasma within the previous 3 months.
* Subject who regularly consumed excessive amounts of alcohol.
* Subject who consumed excessive amount of caffeine (> 5 cups of coffee or equivalent per day).
* Subject who was a smoker (cigarettes and tobacco-related products), or ex-smoker who had smoked in the 3 months preceding the study. Subjects were tested for urinary cotinine at screening.
* Subjects who could not tolerate venepuncture.
* Inability to communicate well with the Investigator (i.e., language problem, poor mental development or impaired cerebral function).
* Participation in a New Chemical Entity clinical study within the previous 4 months or a marketed drug clinical study within the previous 3 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bettica, MD, Study Director — Italfarmaco S.p.A.
Locations (1):
- Simbec Research Ltd, Merthyr Tydfil, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No details are specified in the CSR
Pre-assignment Details: This is a single arm study and not a parallel group study. This means that the participants are 14 in total. The 14 eligible subjects received 1 dose of s.c. Clexane in Treatment Period 1 and 1 dose of S.C. Clexane in Treatment Period 2 (1 dose/period). Each Treatment Period was of 2 days duration.
Groups:
- Clexane 80 mg: Eligible subjects received two doses of s.c. Clexane over 2 Treatment Periods (1 dose/period).
  Each Treatment Period was of 2 days duration, from the afternoon before dosing (Day 0) until 36 hours (h) post-dose (evening of Day 2). Study drug was administered on the morning of Day 1 following an overnight fast.
  There were at least 7 days between each dose administration. In period 1, one dose of Clexane was administered s.c. into the left or right side of the abdomen (alternating sides with Treatment Period). This dose contained 80 mg enoxaparin sodium (equivalent to 8,000 international units (IU) anti-factor Xa (anti FXa activity) in 0.8 mL of water for injection.
  In period 2 one dose of Clexane was administered s.c. into the left or right side of the abdomen (alternating sides with Treatment Period). This dose contained 80 mg enoxaparin sodium (equivalent to 8,000 international units (IU) anti-factor Xa (anti FXa activity) in 0.8 mL of water for injection.
Period: Treatment Period 1
Arm/Group | Clexane 80 mg
Started | 14
Completed (The same 14 subjects received two doses of s.c. Clexane over 2 Treatment Periods (1 dose/period).) | 14
Not Completed | 0
Period: Treatment Period 2
Arm/Group | Clexane 80 mg
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All subjects who received study medication in both Treatment Periods, had sufficient plasma activity/concentration-time profiles and who did not violate the protocol in such a way that may have invalidated or biased the results (major protocol violators) were included in the PK analysis.
Groups:
- Clexane - PK Population: Eligible subjects received two doses of s.c. Clexane over 2 Treatment Periods (1 dose/period).
  Each Treatment Period was of 2 days duration, from the afternoon before dosing (Day 0) until 36 hours (h) post-dose (evening of Day 2). Study drug was administered on the morning of Day 1 following an overnight fast.
  There were at least 7 days between each dose administration. In period 1, one dose of Clexane was administered s.c. into the left or right side of the abdomen (alternating sides with Treatment Period). This dose contained 80 mg enoxaparin sodium (equivalent to 8,000 international units (IU) anti-factor Xa (anti FXa activity) in 0.8 mL of water for injection.
  In period 2 one dose of Clexane was administered s.c. into the left or right side of the abdomen (alternating sides with Treatment Period). This dose contained 80 mg enoxaparin sodium (equivalent to 8,000 international units (IU) anti-factor Xa (anti FXa activity) in 0.8 mL of water for injection.
Arm/Group | Clexane - PK Population
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (8.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Region of Enrollment [Number; unit: participants]
  United Kingdom | 14

OUTCOME MEASURES:

1. Primary Outcome: Anti-FXa Cmax
Description: Enoxaparin exerts its anticoagulant effect primarily via interaction with anti-thrombin III (ATIII), thereby enhancing the inhibitory effect of ATIII on activated factor Xa (FXa) and thrombin/factor IIa (FIIa). Inhibition of FXa activity prevents conversion of prothrombin/factor II (FII) to FIIa and inhibition of FIIa activity (direct/indirect) prevents conversion of fibrinogen to fibrin and therefore clot formation. As enoxaparin cannot be measured directly in blood, the PK of enoxaparin have been studied on the basis of its effect on clotting mechanisms, particularly the inhibition of FXa (anti-FXa) and FIIa (anti-FIIa) activity.
  Cmax is the maximum (or peak) serum concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administered and before the administration of a second dose.
Time Frame: Pre-dose, and at the following times post-dose: 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24 and 36 h in Period 1 and Period 2.
Population: PK Population: All subjects who received study medication in both Treatment Periods, had sufficient plasma activity/concentration-time profiles and who did not violate the protocol in such a way that may have invalidated or biased the results (major protocol violators) were included in the PK analysis.
Measure: Mean (Standard Deviation); unit: IU/mL
Groups:
- Treatment Period 1: Eligible subjects received two doses of s.c. Clexane over 2 Treatment Periods (1 dose/period).
  Each Treatment Period was of 2 days duration, from the afternoon before dosing (Day 0) until 36 hours (h) post-dose (evening of Day 2). Study drug was administered on the morning of Day 1 following an overnight fast.
  There were at least 7 days between each dose administration. In period 1, one dose of Clexane was administered s.c. into the left or right side of the abdomen (alternating sides with Treatment Period). This dose contained 80 mg enoxaparin sodium (equivalent to 8,000 international units (IU) anti-factor Xa (anti FXa activity) in 0.8 mL of water for injection.
- Treatment Period 2: Eligible subjects received two doses of s.c. Clexane over 2 Treatment Periods (1 dose/period).
  Each Treatment Period was of 2 days duration, from the afternoon before dosing (Day 0) until 36 hours (h) post-dose (evening of Day 2). Study drug was administered on the morning of Day 1 following an overnight fast.
  There were at least 7 days between each dose administration. In period 2 one dose of Clexane was administered s.c. into the left or right side of the abdomen (alternating sides with Treatment Period). This dose contained 80 mg enoxaparin sodium (equivalent to 8,000 international units (IU) anti-factor Xa (anti FXa activity) in 0.8 mL of water for injection.
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 14
IU/mL | 0.999 (0.255) | 0.926 (0.204)
Statistical Analysis 1: Comparison: Treatment Period 1 vs Treatment Period 2; Test type: Other — Results were obtained using a mixed-effects ANOVA with fixed effect of study period and a random effect for subject; Geometric least square mean ratio = 93.65, 90% CI 2-sided [87.56 to 100.16]

2. Primary Outcome: Anti-FXa AUC0-t
Description: Enoxaparin exerts its anti-coagulant effect primarily via interaction with anti-thrombin III (ATIII), thereby enhancing the inhibitory effect of ATIII on activated factor Xa (FXa) and thrombin/factor IIa (FIIa). Inhibition of FXa activity prevents conversion of prothrombin/factor II (FII) to FIIa and inhibition of FIIa activity (direct/indirect) prevents conversion of fibrinogen to fibrin and therefore clot formation. As enoxaparin cannot be measured directly in blood, the PK of enoxaparin have been studied on the basis of its effect on clotting mechanisms, particularly the inhibition of FXa (anti-FXa) and FIIa (anti-FIIa) activity.
  AUC0-t is the area under the plasma concentration versus time curve from the time of dosing to the time (t) of the last observed value.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*IU/mL
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 14
h*IU/mL | 9.511 (2.303) | 9.479 (1.990)
Statistical Analysis 1: Comparison: Treatment Period 1 vs Treatment Period 2; Test type: Other — Results were obtained using a mixed-effects ANOVA with fixed effect of study period and a random effect for subject; Geometric least square mean ratio = 100.46, 90% CI 2-sided [95.74 to 105.42]

3. Primary Outcome: Anti-FXa AUC0-inf
Description: Enoxaparin exerts its anti-coagulant effect primarily via interaction with anti-thrombin III (ATIII), thereby enhancing the inhibitory effect of ATIII on activated factor Xa (FXa) and thrombin/factor IIa (FIIa). Inhibition of FXa activity prevents conversion of prothrombin/factor II (FII) to FIIa and inhibition of FIIa activity (direct/indirect) prevents conversion of fibrinogen to fibrin and therefore clot formation. As enoxaparin cannot be measured directly in blood, the PK of enoxaparin have been studied on the basis of its effect on clotting mechanisms, particularly the inhibition of FXa (anti-FXa) and FIIa (anti-FIIa) activity.
  AUC0-inf is the AUC extrapolated to infinity from dosing time, based on the last observed value.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*IU/mL
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 14
h*IU/mL | 9.911 (2.345) | 9.949 (2.050)
Statistical Analysis 1: Comparison: Treatment Period 1 vs Treatment Period 2; Test type: Other — Results were obtained using a mixed-effects ANOVA with fixed effect of study period and a random effect for subject; Geometric least square mean ratio = 101.16, 90% CI 2-sided [96.32 to 106.24]

4. Primary Outcome: Anti-FIIa Cmax
Description: Enoxaparin exerts its anti-coagulant effect primarily via interaction with anti-thrombin III (ATIII), thereby enhancing the inhibitory effect of ATIII on activated factor Xa (FXa) and thrombin/factor IIa (FIIa). Inhibition of FXa activity prevents conversion of prothrombin/factor II (FII) to FIIa and inhibition of FIIa activity (direct/indirect) prevents conversion of fibrinogen to fibrin and therefore clot formation. As enoxaparin cannot be measured directly in blood, the PK of enoxaparin have been studied on the basis of its effect on clotting mechanisms, particularly the inhibition of FXa (anti-FXa) and FIIa (anti-FIIa) activity.
  Cmax is the maximum (or peak) serum concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administered and before the administration of a second dose.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 14
IU/mL | 0.112 (0.027) | 0.107 (0.029)
Statistical Analysis 1: Comparison: Treatment Period 1 vs Treatment Period 2; Test type: Other — Results were obtained using a mixed-effects ANOVA with fixed effect of study period and a random effect for subject; Geometric least square mean ratio = 94.88, 90% CI 2-sided [88.49 to 101.73]

5. Primary Outcome: Anti-FIIA AUC0-t
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*IU/mL
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 14
h*IU/mL | 0.692 (0.233) | 0.696 (0.264)
Statistical Analysis 1: Comparison: Treatment Period 1 vs Treatment Period 2; Test type: Other — Results were obtained using a mixed-effects ANOVA with fixed effect of study period and a random effect for subject; Geometric least square mean ratio = 97.13, 90% CI 2-sided [89.93 to 104.91]

6. Primary Outcome: Anti-FIIA AUC0-inf
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*IU/mL
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 9
h*IU/mL | 1.107 (0.517) | 1.127 (0.366)
Statistical Analysis 1: Comparison: Treatment Period 1 vs Treatment Period 2; Test type: Other — Results were obtained using a mixed-effects ANOVA with fixed effect of study period and a random effect for subject; Geometric least square mean ratio = 108.84, 90% CI 2-sided [95.61 to 123.91]

7. Secondary Outcome: Anti-FXa Tmax
Description: Enoxaparin exerts its anti-coagulant effect primarily via interaction with anti-thrombin III (ATIII), thereby enhancing the inhibitory effect of ATIII on activated factor Xa (FXa) and thrombin/factor IIa (FIIa). Inhibition of FXa activity prevents conversion of prothrombin/factor II (FII) to FIIa and inhibition of FIIa activity (direct/indirect) prevents conversion of fibrinogen to fibrin and therefore clot formation. As enoxaparin cannot be measured directly in blood, the PK of enoxaparin have been studied on the basis of its effect on clotting mechanisms, particularly the inhibition of FXa (anti-FXa) and FIIa (anti-FIIa) activity.
  tmax is the time to Cmax.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 14
hours | 3.50 (0.76) | 4.36 (1.74)

8. Secondary Outcome: Anti-FXa Lambda Zeta
Description: Enoxaparin exerts its anti-coagulant effect primarily via interaction with anti-thrombin III (ATIII), thereby enhancing the inhibitory effect of ATIII on activated factor Xa (FXa) and thrombin/factor IIa (FIIa). Inhibition of FXa activity prevents conversion of prothrombin/factor II (FII) to FIIa and inhibition of FIIa activity (direct/indirect) prevents conversion of fibrinogen to fibrin and therefore clot formation. As enoxaparin cannot be measured directly in blood, the PK of enoxaparin have been studied on the basis of its effect on clotting mechanisms, particularly the inhibition of FXa (anti-FXa) and FIIa (anti-FIIa) activity.
  Lambda zeta is the apparent first-order terminal elimination rate constant calculated from a semi-log plot of the plasma activity/concentration versus time curve.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 14
1/hour | 0.16 (0.06) | 0.14 (0.04)

9. Secondary Outcome: Anti-FXa t1/2
Description: Enoxaparin exerts its anti-coagulant effect primarily via interaction with anti-thrombin III (ATIII), thereby enhancing the inhibitory effect of ATIII on activated factor Xa (FXa) and thrombin/factor IIa (FIIa). Inhibition of FXa activity prevents conversion of prothrombin/factor II (FII) to FIIa and inhibition of FIIa activity (direct/indirect) prevents conversion of fibrinogen to fibrin and therefore clot formation. As enoxaparin cannot be measured directly in blood, the PK of enoxaparin have been studied on the basis of its effect on clotting mechanisms, particularly the inhibition of FXa (anti-FXa) and FIIa (anti-FIIa) activity.
  t1/2 is the apparent first-order terminal elimination half-life calculated as 0.693/kel.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 14
hours | 4.87 (1.39) | 5.19 (1.47)

10. Secondary Outcome: Anti-FXa Cmin
Description: Enoxaparin exerts its anti-coagulant effect primarily via interaction with anti-thrombin III (ATIII), thereby enhancing the inhibitory effect of ATIII on activated factor Xa (FXa) and thrombin/factor IIa (FIIa). Inhibition of FXa activity prevents conversion of prothrombin/factor II (FII) to FIIa and inhibition of FIIa activity (direct/indirect) prevents conversion of fibrinogen to fibrin and therefore clot formation. As enoxaparin cannot be measured directly in blood, the PK of enoxaparin have been studied on the basis of its effect on clotting mechanisms, particularly the inhibition of FXa (anti-FXa) and FIIa (anti-FIIa) activity.
  Cmin is the minimum plasma activity/concentration.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 14
IU/mL | 0.000 (0.0000) | 0.004 (0.0160)

11. Secondary Outcome: Anti-FXa Tmin
Description: Enoxaparin exerts its anti-coagulant effect primarily via interaction with anti-thrombin III (ATIII), thereby enhancing the inhibitory effect of ATIII on activated factor Xa (FXa) and thrombin/factor IIa (FIIa). Inhibition of FXa activity prevents conversion of prothrombin/factor II (FII) to FIIa and inhibition of FIIa activity (direct/indirect) prevents conversion of fibrinogen to fibrin and therefore clot formation. As enoxaparin cannot be measured directly in blood, the PK of enoxaparin have been studied on the basis of its effect on clotting mechanisms, particularly the inhibition of FXa (anti-FXa) and FIIa (anti-FIIa) activity.
  Tmin is time to Cmin. If the minimum value occurred at >1 time point, tmin was defined as the first time point with this value.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 14
hours | 2.57 (9.621) | 0.00 (0.000)

12. Secondary Outcome: Anti-FIIa Tmax
Description: Enoxaparin exerts its anti-coagulant effect primarily via interaction with anti-thrombin III (ATIII), thereby enhancing the inhibitory effect of ATIII on activated factor Xa (FXa) and thrombin/factor IIa (FIIa). Inhibition of FXa activity prevents conversion of prothrombin/factor II (FII) to FIIa and inhibition of FIIa activity (direct/indirect) prevents conversion of fibrinogen to fibrin and therefore clot formation. As enoxaparin cannot be measured directly in blood, the PK of enoxaparin have been studied on the basis of its effect on clotting mechanisms, particularly the inhibition of FXa (anti-FXa) and FIIa (anti-FIIa) activity.
  tmax is time to Cmax. if the maximum value occurred at >1 time point, tmax was defined as the first time point with this value.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 14
hours | 3.61 (0.74) | 4.00 (1.41)

13. Secondary Outcome: Anti-FIIa Lambda Zeta
Description: as for outcome 8
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 9
1/hour | 0.19 (0.08) | 0.17 (0.07)

14. Secondary Outcome: Anti-FIIa t1/2
Description: as for outcome 9
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 9
hours | 4.45 (2.11) | 4.86 (2.02)

15. Secondary Outcome: Anti-FIIa Cmin
Description: as for outcome 10
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 14
IU/mL | 0.000 (0.000) | 0.000 (0.000)

16. Secondary Outcome: Anti-FIIa Tmin
Description: Enoxaparin exerts its anti-coagulant effect primarily via interaction with anti-thrombin III (ATIII), thereby enhancing the inhibitory effect of ATIII on activated factor Xa (FXa) and thrombin/factor IIa (FIIa). Inhibition of FXa activity prevents conversion of prothrombin/factor II (FII) to FIIa and inhibition of FIIa activity (direct/indirect) prevents conversion of fibrinogen to fibrin and therefore clot formation. As enoxaparin cannot be measured directly in blood, the PK of enoxaparin have been studied on the basis of its effect on clotting mechanisms, particularly the inhibition of FXa (anti-FXa) and FIIa (anti-FIIa) activity.
  tmin is the time to minimum concentration.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 14
hours | 0.00 (0.000) | 0.00 (0.000)

17. Secondary Outcome: Thrombin/FIIa Generation AUC0-t
Description: Enoxaparin may have the ability to modulate the fibrinolytic process, by virtue of its ability to inhibit FIIa activity and its generation.
  Thrombin generation test is an integral indicator of the blood clotting system status. This parameter is used for monitoring enoxaparin therapy in patients.
  AUC0-t is the area under the plasma concentration versus time curve from the time of dosing to the time (t) of the last observed value.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*nM
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 14
h*nM | 4034.262 (1955.041) | 4050.840 (1662.359)
Statistical Analysis 1: Comparison: Treatment Period 1 vs Treatment Period 2; Test type: Other — Results were obtained using a mixed-effects ANOVA with fixed effect of study period and a random effect for subject; Geometric least square mean ratio = 102.45, 90% CI 2-sided [96.31 to 109.0]

18. Secondary Outcome: Thrombin/FIIa Generation Cmin
Description: Enoxaparin may have the ability to modulate the fibrinolytic process, by virtue of their ability to inhibit FIIa activity and its generation.
  Thrombin generation test is an integral indicator of the blood clotting system status. This parameter is used for monitoring enoxaparin therapy in patients.
  Cmin is the minimum plasma activity/concentration.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 14
nM | 17.407 (12.562) | 16.971 (12.467)
Statistical Analysis 1: Comparison: Treatment Period 1 vs Treatment Period 2; Test type: Other — Results were obtained using a mixed-effects ANOVA with fixed effect of study period and a random effect for subject; geometric least square mean ratio = 95.84, 90% CI 2-sided [79.11 to 116.11]

19. Secondary Outcome: Thrombin/FIIa Generation Tmin
Description: Enoxaparin may have the ability to modulate the fibrinolytic process, by virtue of its ability to inhibit FIIa activity and its generation.
  Thrombin generation test is an integral indicator of the blood clotting system status. This parameter is used for monitoring enoxaparin therapy in patients.
  Tmin is time to Cmin. If the minimum value occurred at > 1 time-point Tmin was defined as the first time-point with this value.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 14
hours | 3.500 (0.855) | 3.250 (0.803)

20. Secondary Outcome: TFPI Cmax
Description: Enoxaparin also releases tissue factor pathway inhibitor (TFPI), which is thought to contribute to anticoagulant activity, by inhibiting FXa generation and free FXa. Cmax is the maximum (or peak) serum concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administered and before the administration of a second dose.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 14
U/mL | 2.349 (0.464) | 2.344 (0.488)
Statistical Analysis 1: Comparison: Treatment Period 1 vs Treatment Period 2; Test type: Other — Results were obtained using a mixed-effects ANOVA with fixed effect of study period and a random effect for subject; geometric least square mean ratio = 99.54, 90% CI 2-sided [95.69 to 103.54]

21. Secondary Outcome: TFPI Tmax
Description: Enoxaparin also releases tissue factor pathway inhibitor (TFPI), which is thought to contribute to anticoagulant activity, by inhibiting FXa generation and free FXa. Tmax is the time to Cmax. If the maximum value occurred at > 1 time-point Tmax was defined as the first time-point with this value.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 14
hours | 2.79 (2.04) | 2.54 (1.99)

22. Secondary Outcome: TFPI Lambda Zeta
Description: Enoxaparin also releases tissue factor pathway inhibitor (TFPI), which is thought to contribute to anticoagulant activity, by inhibiting FXa generation and free FXa. Lambda zeta is the apparent first-order terminal elimination rate constant calculated from a semi-log plot of the plasma activity/concentration versus time curve. The parameter was calculated by linear least-squares regression analysis using the maximum number of points in the terminal log-linear phase (e.g. ≥ 3 non-zero plasma concentrations).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 6 | 6
1/hour | 0.019 (0.003) | 0.014 (0.005)

23. Secondary Outcome: TFPI T1/2
Description: Enoxaparin also releases tissue factor pathway inhibitor (TFPI), which is thought to contribute to anticoagulant activity, by inhibiting FXa generation and free FXa.
  T1/2 is the apparent first-order terminal elimination half-life calculated as 0.693/kel.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 6 | 6
hours | 37.17 (6.68) | 57.49 (28.92)

24. Secondary Outcome: TFPI AUC0-t
Description: Enoxaparin also releases tissue factor pathway inhibitor (TFPI), which is thought to contribute to anticoagulant activity, by inhibiting FXa generation and free FXa. AUC0-t is the area under the plasma activity/concentration-time curve from the time 0 to the last measurable concentration, as calculated by the linear trapezoidal method.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*U/mL
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 14
h*U/mL | 55.208 (12.282) | 53.937 (9.857)
Statistical Analysis 1: Comparison: Treatment Period 1 vs Treatment Period 2; Test type: Other — Results were obtained using a mixed-effects ANOVA with fixed effect of study period and a random effect for subject; geometric least square mean ratio = 98.36, 90% CI 2-sided [95.31 to 101.51]

25. Secondary Outcome: TFPI AUC0-inf
Description: Enoxaparin also releases tissue factor pathway inhibitor (TFPI), which is thought to contribute to anticoagulant activity, by inhibiting FXa generation and free FXa. AUC0-inf is the area under the activity/concentration-time curve from time 0 extrapolated to infinity. AUC0-inf was calculated as the sum of AUC0-t plus the ratio of the last measurable value to the elimination rate constant.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*U/mL
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 6 | 6
h*U/mL | 123.777 (34.861) | 162.976 (54.363)
Statistical Analysis 1: Comparison: Treatment Period 1 vs Treatment Period 2; Test type: Other — Results were obtained using a mixed-effects ANOVA with fixed effect of study period and a random effect for subject; geometric least square mean ratio = 111.3, 90% CI 2-sided [99.73 to 124.2]

26. Secondary Outcome: TFPI Tmin
Description: Enoxaparin also releases tissue factor pathway inhibitor (TFPI), which is thought to contribute to anticoagulant activity, by inhibiting FXa generation and free FXa. Tmin is the time of Cmin. If the minimum value occurred at > 1 time-point Tmin was defined as the first time-point with this value.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 14
hours | 18.860 (7.263) | 17.430 (5.345)

27. Secondary Outcome: TFPI Cmin
Description: Enoxaparin also releases tissue factor pathway inhibitor (TFPI), which is thought to contribute to anticoagulant activity, by inhibiting FXa generation and free FXa. Cmin is the minimum plasma activity/concentration.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 14
IU/mL | 1.253 (0.291) | 1.227 (0.273)

28. Secondary Outcome: Anti-FXa/Anti-FIIa Cmax
Description: Anti-FXa/anti-FIIa activity Cmax is reported. Cmax is the maximum (or peak) serum concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administered and before the administration of a second dose.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 14
U/mL | 9.095 (1.464) | 9.020 (1.838)
Statistical Analysis 1: Comparison: Treatment Period 1 vs Treatment Period 2; Test type: Other — Results were obtained using a mixed-effects ANOVA with fixed effect of study period and a random effect for subject; geometric least square mean ratio = 98.7, 90% CI 2-sided [93.16 to 104.57]

29. Secondary Outcome: Anti-FXa/Anti-FIIa AUC0-t
Description: Anti-FXa/anti-FIIa activity AUC0-t is reported. AUC0-t is the area under the plasma activity/concentration-time curve from the time 0 to the last measurable concentration, as calculated by the linear trapezoidal method.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*nM
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 14
h*nM | 15.137 (5.619) | 16.927 (12.466)
Statistical Analysis 1: Comparison: Treatment Period 1 vs Treatment Period 2; Test type: Other; geometric least square mean ratio = 103.43, 90% CI 2-sided [94.5 to 113.2]

30. Secondary Outcome: Anti-FXa/Anti-FIIa AUC0-inf
Description: Anti-FXa/anti-FIIa activity AUC0-inf is reported. AUC0-inf is the AUC extrapolated to infinity from dosing time, based on the last observed value.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*U/mL
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 9
h*U/mL | 10.143 (3.184) | 8.941 (2.545)
Statistical Analysis 1: Comparison: Treatment Period 1 vs Treatment Period 2; Test type: Other; geometric least square mean ratio = 92.92, 90% CI 2-sided [80.58 to 107.16]

31. Secondary Outcome: Anti-FXa/Anti-FIIa Tmax
Description: Anti-FXa/anti-FIIa activity Tmax is reported. Tmax is the Time to Cmax. If the maximum value occurred at > 1 time-point Tmax was defined as the first time-point with this value.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 14
hours | 1.02 (0.33) | 1.11 (0.33)

32. Secondary Outcome: Anti-FXa/Anti-FIIa Lambda Zeta
Description: Anti-FXa/anti-FIIa activity lambda zeta is reported. Lambda zeta is the apparent first-order terminal elimination rate constant calculated from a semi-log plot of the plasma activity/concentration versus time curve. The parameter was calculated by linear least-squares regression analysis using the maximum number of points in the terminal log-linear phase (e.g. ≥ 3 non-zero plasma concentrations).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 9
1/hour | 1.09 (0.91) | 1.05 (0.58)

33. Secondary Outcome: Anti-FXa/Anti-FIIa t1/2
Description: Anti-FXa/anti-FIIa activity t1/2 is reported. t1/2 is the apparent first-order terminal elimination half-life calculated as 0.693/kel.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 9
hours | 1.37 (0.80) | 1.30 (0.81)

34. Secondary Outcome: Number of Patients With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs and Severity of TEAEs
Description: Description of adverse event profile in healthy volunteers after administration of Enoxaparin sodium s.c. as above described.
Time Frame: as for outcome 1
Population: Safety Population: All subjects who received at least 1 dose of study medication were included in the safety analysis.
Measure: Number; unit: participants
Arm/Group | Treatment Period 1 | Treatment Period 2
Number analyzed (Participants) | 14 | 14
participants
  TEAEs | 4 | 2
  serious TEAEs | 0 | 0
  TEAEs heading to withdrawal | 0 | 0
  Mild TEAEs | 3 | 2
  Moderate TEAEs | 1 | 0
  TEAEs not related | 1 | 1
  TEAEs related | 2 | 1
  TEAEs Unkown | 1 | 0

ADVERSE EVENTS:
Time Frame: At Day 0, 1 and 2 during treatment period 1, and Day 0, 1 and 2 during treatment period 2.
Arm/Group | Treatment Period 1 | Treatment Period 2
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 4/14 | 2/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Period 1 (N=14) | Treatment Period 2 (N=14)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No